CLINICAL TRIAL: NCT01588405
Title: A Multicenter, Open-Label Study of the Safety and Tolerability of Transitioning From Remodulin® to Oral Treprostinil in Subjects With Pulmonary Arterial Hypertension
Brief Title: Remodulin® to Oral Treprostinil Transition
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: United Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TDE-PH-205
Record Dates: First submitted 2012-01-06; First posted 2012-05-01 (Estimated); Results first posted 2016-05-16 (Estimated); Last update posted 2016-05-16 (Estimated); Status verified 2016-04

CONDITIONS: Pulmonary Arterial Hypertension
Keywords: Pulmonary Arterial Hypertension; UT-15C SR; PAH
MeSH Terms: conditions — Pulmonary Arterial Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- UT-15C SR (Experimental)
  Interventions: Drug: UT-15C SR

INTERVENTIONS:
Drug: UT-15C SR — Subjects will transition in the hospital from Remodulin to UT-15C SR within 5 days of the start of the transition. The dose of Remodulin will be decreased as the dose of UT-15C SR is increased over the 5 days. Once subjects have been transitioned from Remodulin, the dose of UT-15C SR will continue to be modified / titrated to the appropriate optimal dose for that subject throughout the rest of the study.

SUMMARY:
This multi-center, open-label study will assess the tolerability and safety of transitioning subjects with stable Pulmonary Arterial Hypertension (PAH) from continuous intravenous (IV) or subcutaneous (SC) Remodulin infusion to oral treprostinil (UT-15C sustained release (SR) tablets).

This study will consist of an in-hospital transition phase, dose optimization/evaluation phase, and follow up phase.

ELIGIBILITY:
Inclusion Criteria:

* Between 15 and 80 years of age, inclusive, weigh at least 40 kg and have a diagnosis of PAH
* Have stable disease as confirmed by recent right heart catheterization and a Baseline 6MWD of at least 250 meters
* Have been receiving Remodulin for at least 90 days and at a stable dose for at least 30 days prior to the Baseline visit; the dose of Remodulin must be between 25-75 ng/kg/min, inclusive
* Must be also receiving an endothelin receptor antagonist (ERA) and/or a phosphodiesterase-5 inhibitor (PDE-5i) for at least 90 days and have been at a stable dose for at least 30 days prior to Baseline

Exclusion Criteria:

* WHO functional class III and IV subjects will be excluded

Ages: 15 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2012-04; Primary Completion 2014-07 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia Madden, MD, MPH, Study Chair — Senior Clinical Research Physician
Locations (6):
- United States (6):
  - Arizona Pulmonary Specialists, Phoenix, Arizona
  - University of Arizona Clinical and Translational Science (CATS) Research Center, Tucson, Arizona
  - Washington University School of Medicine, St Louis, Missouri
  - University of Rochester, Rochester, New York
  - The Ohio State University, Columbus, Ohio
  - University of Pittsburgh Medical Center (UPMC), Pittsburgh, Pennsylvania

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | UT-15C SR
Started | 33
Completed | 31
Not Completed | 2
Not completed — Adverse Event | 1
Not completed — Clinical Worsening | 1

BASELINE CHARACTERISTICS:
Arm/Group | UT-15C SR
Number analyzed (Participants) | 33
Age, Continuous [Median (Full Range); unit: years] | 50.0 [18 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25
  Male | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 1
  White | 28
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants That Were Succesfully Transitioned From Parenteral Remodulin to UT-15C.
Description: Successful transition was based on the number of participants that completely transitioned to oral treprostinil by the week 4 study visit and clinically maintained on oral treprostinil treatment through Week 24.
Time Frame: Up to 24 weeks
Measure: Number; unit: participants
Arm/Group | UT-15C SR
Number analyzed (Participants) | 33
participants | 31

2. Secondary Outcome: Change From Baseline in Six-minute Walk Distance at Week 24
Description: The purpose of the 6MWT is to evaluate exercise capacity associated with carrying out activities of daily living. Patients were instructed to walk down a corridor at a comfortable speed as far as they could manage for six minutes, resting whenever they needed. Distance <500 meters suggests considerable exercise limitation; Distance 500-800 meters suggests moderate limitation; Distance >800 meters (with no rests) suggests mild or no limitation.
Time Frame: Baseline and week 24
Population: One subject completed the Week 24 visit but was unable to undergo all assessments. As such, the evaluable data at Week 24 was summarized mainly using an N of 30 subjects.
Measure: Median (Full Range); unit: meters
Arm/Group | UT-15C SR
Number analyzed (Participants) | 30
meters
  6MWD at Week 24 | 467 [305 to 715]
  6MWD Change from Baseline | 16.7 [-98.0 to 95.0]

3. Secondary Outcome: Change in Borg Dyspnea Score (Following 6MWT) From Baseline to Week 24
Description: The Borg dyspnea score is a 10-point scale rating the maximum level of dyspnea (difficulty in breathing) experienced during the six-minute walk test (6MWT). The Borg dyspnea score was assessed immediately following the 6MWT. Scores ranged from 0 (for no shortness of breath) to 10 (for the greatest shortness of breath ever experienced).
Time Frame: Baseline and week 24
Population: as for outcome 2
Measure: Median (Full Range); unit: units on a scale
Arm/Group | UT-15C SR
Number analyzed (Participants) | 30
units on a scale | 0.0 [-3.5 to 3.0]

4. Secondary Outcome: Change in Quality of Life (QoL) Assessment: Cambridge Pulmonary Hypertension Outcome Review (CAMPHOR) From Baseline to Week 24
Description: The CAMPHOR is a health related quality of life instrument validated for pulmonary hypertension that assesses impairment (symptoms), disability (activities) and quality of life. The questionnaire is divided into three sections; Symptoms (Scores 0-25; high scores indicate more symptoms), Activity (Score 0-30; low score indicates good functioning) and Quality of Life (0-25; high scores indicate poor QoL). The sum of these scores equates to the Total score (0-80). In the CAMPHOR scores, lower scores indicate improvements.
Time Frame: Baseline and week 24
Measure: Median (Full Range); unit: units on a scale
Arm/Group | UT-15C SR
Number analyzed (Participants) | 31
units on a scale
  Symptom | -1.0 [-11 to 7]
  Activity | 0.0 [-8 to 8]
  Quality of Life | 0.0 [-14 to 3]
  Total Camphor Score | -2.0 [-25 to 17]

5. Secondary Outcome: Change in World Health Organization (WHO) Functional Classification From Baseline to Week 24
Description: Class I: No limitation of physical activity. Class II: Slight limitation of physical activity. Class III: Marked limitation of physical activity. Class IV: Inability to carry out any physical activity without symptoms.
Time Frame: Baseline and Week 24
Population: The World Health Organization (WHO) Functional Classification was only conducted at baseline for one subject, because the subject discontinued the study prior to the collection of this assessment at the next visit. One subject had this assessment prior to study discontinuation.
Measure: Number; unit: participants
Arm/Group | UT-15C SR
Number analyzed (Participants) | 32
participants
  I to I | 3
  I to II | 2
  I to III | 1
  II to I | 3
  II to II | 21
  II to III | 1
  Missing | 1

6. Secondary Outcome: Change in Dyspnea-fatigue Index From Baseline to Week 24
Description: The dyspnea-fatigue index has three components, each rated on a scale of 0 to 4, for the magnitude of the task that evokes dyspnea or fatigue, the magnitude of the pace (or effort) with which the task is performed and the associated functional impairment in general activities. The ratings for each component were added to form an aggregate score, which could range from 0, for the worst condition, to 12, for the best.
Time Frame: Baseline and Week 24
Measure: Median (Full Range); unit: units on a scale
Arm/Group | UT-15C SR
Number analyzed (Participants) | 31
units on a scale | 1.0 [-3 to 4]

7. Secondary Outcome: Change From Baseline to Week 24 in Pharmacokinetic Parameters: Peak Plasma Concentration (Cmax), Average Plasma Concentration (Cavg), and Trough Plasma Concentration (Cmin)
Description: Treprostinil pharmacokinetics (PK) were evaluated on two occasions during this study, once while the subject was still receiving Remodulin and again at Week 24 when the subject was receiving a stable dose of oral treprostinil. Blood samples were scheduled to be drawn from each subject initially at time 0 and the following subsequent times: 2, 4, 5, 6, 8, 10 and 12 hours after time of study drug administration (time 0) for a total of eight samples.
Time Frame: Baseline and Week 24
Population: Dosing frequency was modified for BID to TID during the study, reported separately for patients on BID vs TID dosing at week 24. The number of participants analyzed is inconsistent with participant flow because it includes data from an early termination patient. A pharmacokinetics sample collected at early termination was included in the analysis.
Measure: Median (Full Range); unit: (ng/mL)
Groups:
- IV Remodulin / SQ Remodulin: Baseline while on infused Remodulin
- UT-15C SR (BID): Subjects who were on BID dosing of UT-15C SR at week 24
- UT-15C SR (TID): Subjects who were on TID dosing of UT-15C SR at week 24
Arm/Group | IV Remodulin / SQ Remodulin | UT-15C SR (BID) | UT-15C SR (TID)
Number analyzed (Participants) | 32 | 6 | 26
(ng/mL)
  Cmax (ng/mL) | 8.76 [3.91 to 20.9] | 13 [9.41 to 20.8] | 12.1 [0.899 to 38.9]
  Cavg (ng/mL) | 7.22 [2.85 to 15.4] | 6.89 [4.26 to 11.2] | 6.64 [0.345 to 22.6]
  Cmin (ng/mL) | 5.63 [2.09 to 11.9] | 1.94 [1.30 to 2.97] | 2.45 [0.0489 to 18.6]

8. Secondary Outcome: Change From Baseline to Week 24 in Pharmacokinetics Parameter: Peak Time to Reach Peak Plasma Concentration [Tmax (h)]
Description: as for outcome 7
Time Frame: Baseline and Week 24
Population: as for outcome 7
Measure: Mean (Full Range); unit: [Tmax (h)]
Arm/Group | IV Remodulin / SQ Remodulin | UT-15C SR (BID) | UT-15C SR (TID)
Number analyzed (Participants) | 32 | 6 | 26
[Tmax (h)] | 4.01 [0.00 to 12.00] | 5.60 [3.98 to 6.0] | 3.92 [0.00 to 8.17]

9. Secondary Outcome: Change From Baseline to Week 24 in Pharmacokinetics Parameters: Area Under the Plasma Concentration Curve (AUC) [h(ng/mL)]
Description: as for outcome 7
Time Frame: Baseline and Week 24
Population: The number of participants analyzed is inconsistent with participant flow because it includes data from an early termination patient. A pharmacokinetics sample collected at early termination was included in the analysis.
Measure: Median (Full Range); unit: [h(ng/mL)]
Arm/Group | IV Remodulin / SQ Remodulin | UT-15C SR (BID) | UT-15C SR (TID)
Number analyzed (Participants) | 32 | 6 | 26
[h(ng/mL)] | 86.3 [34.2 to 185] | 82.5 [49.7 to 134] | 81.8 [7.18 to 277]

10. Secondary Outcome: Change From Baseline to Week 24 in Hemodynamics Parameters: Mean Pulmonary Artery Pressure (PAPm), Mean Right Atrial Pressure (RAPm) and Mean Pulmonary Capillary Wedge Pressure (PCWPm)
Description: Pulmonary hypertension (PH) is an increase in pressure in the pulmonary vasculature defined as a mean pulmonary artery pressure (PAPm) greater than 25 mmHg at rest or greater than 30 mmHg with exercise, as measured by right heart catheterization. Right Atrial Pressure (RAP) is the pressure of blood in the right atrium of the heart. Pulmonary Capillary Wedge Pressure (PCWP) is used to calculated pulmonary vascular resistance and can help guide therapeutic efficacy. The PAPm, RAPm and PCWPm values and their respective changes from Baseline to Week 24 at peak exercise were measured by Swan-Ganz right heart catheterization.
Time Frame: Baseline and week 24
Population: One subject completed the Week 24 visit but was unable to undergo these assessments. As such, the evaluable data at Week 24 was summarized using an N of 30 subjects, which is why the number of participants analyzed is inconsistent with the participant flow module.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | UT-15C SR
Number analyzed (Participants) | 30
mmHg
  PAPm (mmHg) | 2.2 (8.6)
  RAPm (mmHg) | 0.5 (3.7)
  PCWPm (mmHg) | 0.6 (4.6)

11. Secondary Outcome: Change From Baseline to Week 24 in Hemodynamics Parameters: Arterial Oxygen Saturation (SaO2) (%) and Mixed Venous Oxygen Saturation (SvO2) (%)
Description: SaO2 measured by Arterial Blood Draw and Blood Gas Analyzer and SvO2 measured via Pulmonary Artery Catheter, are both Hemodynamics Parameters collected during right heart catheterization. Mixed venous oxygen saturation (SvO2) can help to determine whether the cardiac output and oxygen delivery is high enough to meet a patient's needs
Time Frame: Baseline and Week 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percent of Oxygen saturation
Arm/Group | UT-15C SR
Number analyzed (Participants) | 30
Percent of Oxygen saturation
  SaO2 (%) | -0.1 (3.4)
  SvO2 (%) | -3.2 (5.2)

12. Secondary Outcome: Change From Baseline to Week 24 in Hemodynamics Parameters: Cardiac Output (CO) (L/Min)
Description: Cardiac Output (CO) is the volume of blood ejected by the heart per minute, as measured by right heart catheterization. The value and change from Baseline to Week 24 at peak exercise was measured by Swan-Ganz right heart catheterization.
Time Frame: Baseline and week 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: L/min
Arm/Group | UT-15C SR
Number analyzed (Participants) | 30
L/min | -0.3 (1.3)

13. Secondary Outcome: Change From Baseline to Week 24 in Hemodynamics Parameters: Cardiac Index (CI) (L/Min/m^2)
Description: Cardiac Index (CI) relates the cardiac output (CO) from left ventricle to body surface area (BSA), thus relating heart performance to the size of the individual. The CI values and their respective changes from Baseline to Week 24 at peak exercise was measured by Swan-Ganz right heart catheterization.
Time Frame: Baseline and week 24
Population: Both the Thermodilution (n=6) and Fick (n=29) methods were used to determine CO and in some cases both methods were utilized; however, only the Fick method was used for (CI) for the purpose of this analysis and included only 29 subjects.
Measure: Mean (Standard Deviation); unit: L/min/m^2
Arm/Group | UT-15C SR
Number analyzed (Participants) | 29
L/min/m^2 | -0.1 (0.7)

14. Secondary Outcome: Change From Baseline to Week 24 in Hemodynamics Parameters: Pulmonary Vascular Resistance Index (PVRI) (mmHg*Min*m^2/L)
Description: Pulmonary Vascular Resistance Index (PVRI) is calculated using Mean Pulmonary Arterial Pressure(PAPm), Pulmonary Capillary Wedge Pressure (PCWP) and Cardiac Index (CI ), to provide information about right ventricular overload. The PVRI values and their respective changes from Baseline to Week 24 at peak exercise was measured by Swan-Ganz right heart catheterization.
Time Frame: Baseline and week 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mmHg*min*m^2/L
Arm/Group | UT-15C SR
Number analyzed (Participants) | 30
mmHg*min*m^2/L | 1.6 (4.8)

15. Secondary Outcome: Change From Baseline to Week 24 in Hemodynamics Parameters: Pulmonary Vascular Resistance (PVR) (mmHg*Min/L)
Description: pulmonary vascular resistance (PVR) is the resistance the right ventricle must overcome to pump blood into the pulmonary arteries. The change in PVR values from Baseline to Week 24 at peak exercise were measured by Swan-Ganz right heart catheterization.
Time Frame: Baseline and week 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mmHg*min/L
Arm/Group | UT-15C SR
Number analyzed (Participants) | 30
mmHg*min/L | 0.8 (2.4)

ADVERSE EVENTS:
Time Frame: Adverse events were recorded throughout the 24-week study, including the screening and follow-up phase, as well as 30 days post end of study visit.
Arm/Group | UT-15C SR
Serious Adverse Events (participants affected / at risk) | 9/33
Other Adverse Events (participants affected / at risk) | 32/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | UT-15C SR (N=33)
Diarrhoea (Gastrointestinal disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 2 (2)
Vertigo (Nervous system disorders) | 2 (2)
Abdominal Distension (Gastrointestinal disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Ascites (Hepatobiliary disorders) | 1 (1)
Atrial Flutter (Cardiac disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Gastric Ulcer (Gastrointestinal disorders) | 1 (1)
Gastroenteritis Viral (Infections and infestations) | 1 (1)
Lung carcinoma cell type unspecified stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1)
Pleurisy (Cardiac disorders) | 1 (1)
Renal Failure Acute (Renal and urinary disorders) | 1 (1)
Systemic Lupus Erythematosus (Immune system disorders) | 1 (1)
Ventricular Extrasystoles (Cardiac disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Chronic Hepatic Failure (Hepatobiliary disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | UT-15C SR (N=33)
Headache (Nervous system disorders) | 28 (29)
Nausea (Gastrointestinal disorders) | 22 (26)
Flushing (Vascular disorders) | 23 (28)
Diarrhoea (Gastrointestinal disorders) | 20 (23)
Fatigue (General disorders) | 16 (16)
Vomiting (Gastrointestinal disorders) | 14 (19)
Dyspepsia (Gastrointestinal disorders) | 13 (13)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 9 (12)
Upper Resipiratory Tract Infection (Respiratory, thoracic and mediastinal disorders) | 10 (12)
Dizziness (Nervous system disorders) | 8 (10)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 8 (8)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 8 (8)
Fluid Retention (Metabolism and nutrition disorders) | 6 (7)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 6 (6)
Abdominal distension (Gastrointestinal disorders) | 4 (6)
Abdominal Pain (Gastrointestinal disorders) | 5 (5)
Back Pain (Musculoskeletal and connective tissue disorders) | 5 (5)
Palpitations (Cardiac disorders) | 4 (4)
Tachycardia (Cardiac disorders) | 5 (5)
Constipation (Gastrointestinal disorders) | 4 (4)
Insomnia (Psychiatric disorders) | 4 (4)
Edema Peripheral (Eye disorders) | 4 (5)
Rash (Skin and subcutaneous tissue disorders) | 4 (5)
Anxiety (Psychiatric disorders) | 3 (3)
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Nasopharyngitis (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Pain (General disorders) | 3 (3)
Renal Failure Acute (Renal and urinary disorders) | 3 (4)
Weight Decreased (Investigations) | 3 (3)
Weight Increased (Investigations) | 3 (3)
Decreased Appetite (Metabolism and nutrition disorders) | 3 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (3)
Chest Discomfort (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Chills (General disorders) | 2 (2)
Dermatitis (Skin and subcutaneous tissue disorders) | 2 (2)
Dry Mouth (General disorders) | 2 (2)
Dyspnea Exertional (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Epistaxis (Vascular disorders) | 2 (2)
Gastroenteritis (Gastrointestinal disorders) | 2 (2)
Hypotension (Vascular disorders) | 2 (3)
Iron Deficiency Anemia (Blood and lymphatic system disorders) | 2 (2)
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 2 (2)
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Ocular hyperemia (Eye disorders) | 2 (2)
Pyrexia (General disorders) | 2 (2)
Rectal Hemorrhage (Gastrointestinal disorders) | 2 (2)
Rhinitis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Sinusitis (Immune system disorders) | 2 (3)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institution and/or Principal Investigator agree not to publish or publicly present any interim results of the Study without the prior written consent of Sponsor, not to be unreasonably withheld or delayed, except as provided below. Institution and/or Principal Investigator further agree to provide Sponsor with drafts of any such publication or presentation for review and approval no less than 30 days prior to submission for publication or the date of public presentation.